CLINICAL TRIAL: NCT07264569
Title: Phase Ib/II Clinical Study to Evaluate the Safety, Tolerability, Biodistribution Characteristics and Preliminary Efficacy of BioTTT001 in the Treatment of Patients With Recurrent/Progressive Non-small Cell Lung Cancer
Brief Title: Evaluate the Safety, Tolerability, Biodistribution Characteristics and Preliminary Efficacy of BioTTT001
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HXNY-BM-01
Record Dates: First submitted 2025-05-19; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2024-12

CONDITIONS: Meningeal Metastasis
MeSH Terms: conditions — Meningeal Carcinomatosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recombinant human nsIL12 oncolytic adenovirus injection( BioTTT001 injection) (Experimental): BioTTT001 is administered as a Intrathecal injection using an Ommaya reservoir.The dosage administered to the subjects is determined based on the group they belong to. This study establishes three dosage groups: 1.0×10^9 VP, 5.0×10^9 VP, and 1.0×10^10 VP.In the first week, the drug is administered 3 times, followed by 1 dose every 3 weeks thereafter. In the phase Ib dose escalation study, participants can receive up to 6 doses, while in the phase II dose expansion study, participants will be treated until disease progression (PD), intolerable toxicity, the start of new anti-tumor treatment, termination of treatment decided upon careful consideration by the participant or investigator, death, or loss to follow-up (whichever occurs first).
  Interventions: Biological: BioTTT001 injection

INTERVENTIONS:
Biological: BioTTT001 injection — BioTTT001 is administered as a Intrathecal injection using an Ommaya reservoir.The dosage administered to the subjects is determined based on the group they belong to. This study establishes three dosage groups: 1.0×10^9 VP, 5.0×10^9 VP, and 1.0×10^10 VP.

SUMMARY:
Phase Ib/II clinical study on evaluating the safety, tolerance, biodistribution characteristics and preliminary efficacy of recombinant human nsIL12 oncolytic adenovirus injection (BioTT001) in the treatment of meningeal metastasis in recurrent/progressive non-small cell lung cancer

DETAILED DESCRIPTION:
This study is a single-arm, open-label, dose-escalation and dose-expansion phase Ib/II clinical trial aimed at evaluating the safety, tolerability, biological distribution characteristics, and preliminary efficacy of recombinant human nsIL12 oncolytic adenovirus injection (BioTTT001) in patients with recurrent/progressive non-small cell lung cancer with meningeal metastases. The study is divided into two phases: the phase Ib dose-escalation .The dose escalation phase establishes three dosage groups, namely 1.0×10^9 VP, 5.0×10^9 VP, and 1.0×10^10 VP and the phase II dose-expansion.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 70 years old (including boundary values);
2. Patients diagnosed with NSCLC through pathological histology, who have experienced recurrence or progression after standard treatment, and have tumor cells found in cerebrospinal fluid or MRI diagnosis of leptomeningeal metastasis;
3. Performance Status (PS) score ≤ 3 points;
4. Suitable for Ommaya reservoir placement as determined by the investigator, and meet the conditions for drug administration;
5. Expected survival ≥ 3 months;
6. Good organ function, defined as follows:

   1. Blood routine (not having received blood transfusion or other treatments within 14 days): Absolute neutrophil count ≥ 1.5 × 10^9/L, platelet count ≥ 100 × 10^9/L, hemoglobin ≥ 90 g/L, white blood cell count ≥ 3.0 × 10^9/L;
   2. Coagulation function: Activated Partial Thromboplastin Time (APTT) ≤ 1.5 times the upper limit of normal (ULN), International Normalized Ratio (INR) ≤ 1.5 times ULN;
   3. Liver function: Total bilirubin (TBIL) ≤ 1.5 times ULN, Gilbert's syndrome participants should be ≤ 3 times ULN, Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤ 3 times ULN (if there is liver metastasis, ALT or AST ≤ 5 times ULN);
   4. Renal function: Serum creatinine ≤ 1.5 times ULN, or creatinine clearance rate ≥ 50 mL/min (Cockcroft-Gault formula calculation see Appendix 3);
7. Voluntarily participate and sign the informed consent form after being explained the study content before the start of the relevant procedures;
8. For participants and partners with reproductive capacity and sexual activity, must agree to use medically approved effective contraception methods during treatment and for 6 months after the last dose, such as double-barrier contraception, and men agree not to donate sperm;
9. For women with reproductive capacity, the blood pregnancy test result within 7 days before the first dose must be negative, and willing to undergo additional pregnancy tests during the study. Reproductive capacity refers to women who have not undergone surgical sterilization (i.e., bilateral tubal ligation, bilateral oophorectomy, or total hysterectomy) or are not postmenopausal; Menopause is defined as amenorrhea ≥ 12 months in women over 45 years old, excluding other causes of amenorrhea. Additionally, for women under 50 years old, serum Follicle-Stimulating Hormone (FSH) levels must be in the postmenopausal range to confirm menopause;
10. Good compliance, willing and able to follow all study procedures and cooperate with observation and follow-up.
11. If patients have previously received tyrosine kinase inhibitors (TKIs) treatment for more than two weeks and have only brain progression, they should continue the TKIs treatment during the enrollment period and cannot arbitrarily switch to other TKIs.

Exclusion Criteria:

1. Patients who have received systemic antitumor therapy within two weeks, including intravenous chemotherapy, intrathecal chemotherapy, or whole-brain radiotherapy (excluding immunotherapy);
2. immunotherapy administered within 6 weeks prior to the first dose;
3. traditional Chinese medicine with antitumor indications administered within 2 weeks prior to the first dose;
4. patients with uncontrolled epilepsy;
5. those who received any other investigational drug within 4 weeks prior to the first dose;
6. major organ surgeries (excluding biopsy) or significant trauma within 4 weeks prior to the first dose, or those requiring elective surgery during the study;
7. patients with prior history of cell therapy, gene therapy, or oncolytic virus therapy;
8. individuals with known or suspected allergies to active ingredients, excipients, or contrast agents in the study drug or imaging contrast agents;
9. patients with organ transplant history or planned organ transplant during the study;
10. active infections requiring systemic intravenous treatment or uncontrolled infections, or unexplained fever>38.5℃ occurring during screening or before the first dose;
11. patients with severe coagulation disorders or evidence of significant bleeding risk; history of gastrointestinal bleeding; any other CTCAE 2-level or higher bleeding events within 6 months;
12. participants who received immunosuppressants (e.g., azathioprine, cyclophosphamide, methotrexate, thalidomide) within 14 days prior to the first dose;
13. patients whose adverse reactions from previous antitumor therapy have not resolved to a CTCAE 5.0 grade ≤1 (excluding non-safety-related toxicities like alopecia as determined by investigators);
14. patients with immunodeficiency history, including HIV antibody-positive status;
15. Active hepatitis B (HBsAg-positive with HBV-DNA> 500 IU/mL or laboratory test lower limit [only when the laboratory test lower limit exceeds 500 IU/mL]); Active hepatitis C (HCV antibody positive with HCV-RNA> laboratory test lower limit); Positive Treponema pallidum antibody;
16. Hypertension poorly controlled by investigators (uncontrolled arterial hypertension despite standardized treatment: systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥100 mmHg);
17. History of severe cardiovascular disease: such as clinically managed ventricular arrhythmias; QTc interval> 480 ms; Acute coronary syndrome, congestive heart failure, stroke, or other Grade III or higher cardiovascular events within 6 months prior to first dose; New York Heart Association (NYHA) class II or left ventricular ejection fraction (LVEF) <50%;
18. Concurrent presence of other uncured malignancies within 3 years (excluding clinically curable precancerous conditions like cervical carcinoma in situ and basal cell carcinoma);
19. Active or recurrent autoimmune diseases (including but not limited to systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.) except clinically stable autoimmune thyroiditis;
20. Vaccination history within 4 weeks prior to first dose (live attenuated vaccines/recombinant vaccines) or within 2 weeks prior to first dose (inactivated vaccines);
21. Previous immunotherapy with irAE grade ≥3;
22. Patients with intracranial brainstem metastases or rapidly progressing diffuse cerebral parenchymal metastases;
23. those showing tumor enhancement margins invading ventricular walls on cranial MRI or postoperative ventricular communication;
24. history of encephalitis, multiple sclerosis, or other CNS infections;
25. cerebral herniation syndrome;
26. confirmed alcohol/drug dependence;
27. psychiatric disorders or poor compliance;
28. Pregnant or lactating women;
29. Researchers believe that due to other serious systemic diseases or other reasons, the subjects are not suitable to participate in this clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
DLT, MTD and/or RP2D | Progress-free survival time
  DLT, MTD and/or RP2D
Phase Ib dose-escalation study | 28 days within BioTTT001 injection
  DLT, MTD and/or RP2D;The incidence and severity of adverse events (AE) assessed based on the NCI CTCAE Version 5.0 standard.

CONTACTS AND LOCATIONS:
Locations (1):
- Phase Ib/II Clinical Study to Evaluate the Safety, Tolerability, Biodistribution Characteristics and Preliminary Efficacy of Recombinant Human nsIL12 Oncolytic Adenovirus Injection (BioTTT001) in the Treatment of Patients With Recurrent/Progressive Non-s, Zhengzhou, Henan, China